CLINICAL TRIAL: NCT01821612
Title: Neoadjuvant FOLFIRINOX and Chemoradiation Followed by Definitive Surgery and Postoperative Gemcitabine for Patients with Borderline Resectable Pancreatic Adenocarcinoma: an Intergroup Single-Arm Pilot Study
Brief Title: Chemotherapy and Radiation Therapy Before Surgery Followed by Gemcitabine in Treating Patients with Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A021101; U10CA031946 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Capecitabine; Radiation; Surgical Procedures, Operative; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mFOLFIRINOX, chemoradiation, surgery and gemcitabine (Other): Each patient will receive mFOLFIRINOX therapy administered every other week for a total of 4 cycles. Each treatment cycle is a total of 14 days. This treatment program consists of four drugs (oxaliplatin 85 mg/m^2 IV over 2 hours on day 1 followed by irinotecan 180 mg/m^2 IV over 90 minutes on day 1 followed by, leucovorin 400 mg/m^2 IV over 2 hours on day 1 followed by 5-FU 2400 mg/m^2 IV over 46-48 hours).
  Two to six weeks following treatment with the mFOLFIRINOX, if the tumor has not spread to other parts of the body then the patient will receive capecitabine 825 mg/m^2, twice daily for 28 days along with radiation therapy. Patients will have surgery within 4-10 weeks of the last dose of chemoradiation if the tumor has gotten smaller or stayed the same.
  Within 6-8 weeks following surgery, patients will receive gemcitabine for 2 cycles (1 cycle is 28 days). Gemcitabine will be given IV on days 1, 8 and 15 of every 28 day cycle.
  Interventions: Drug: oxaliplatin; Drug: irinotecan; Drug: leucovorin; Drug: 5-fluorouracil; Drug: capecitabine; Radiation: radiation; Procedure: surgery; Drug: gemcitabine

INTERVENTIONS:
Drug: oxaliplatin — IV
Drug: irinotecan — IV
Drug: leucovorin — IV
Drug: 5-fluorouracil — IV
Drug: capecitabine — PO
Radiation: radiation
Procedure: surgery
Drug: gemcitabine — IV

SUMMARY:
This pilot clinical trial studies combination chemotherapy and radiation therapy before surgery followed by gemcitabine hydrochloride in treating patients with pancreatic cancer. Drugs used in chemotherapy, such as oxaliplatin, irinotecan hydrochloride, leucovorin calcium, fluorouracil, and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new treatment program for patients with borderline resectable pancreas cancer in order to determine what effects, good and bad, chemotherapy and chemoradiation have on your cancer and to see if it allows safe surgery.

Primary Objectives:

* To assess the accrual rate of this study.
* To assess the rate of treatment-related toxicity and treatment delay during preoperative therapy.
* To assess the rate of completion of all preoperative and operative therapy.

Secondary Objectives:

* To assess the macroscopic (R0/R1) resection rate.
* To estimate the rate of radiographic and histopathologic response to preoperative therapy.
* To estimate the time to locoregional and distant recurrence.
* To assess overall survival (OS).
* To retrieve nucleic acids from pretreatment pancreatic ductal adenocarcinoma biopsies and to assess the quality of these nucleic acids using a sequencing-based assessment of tumor DNA.

ELIGIBILITY:
Pre-Registration Eligibility Criteria

* Documentation of Disease and Radiographic Staging

  * Cytologic or histologic proof of adenocarcinoma of the pancreatic head or uncinate process
  * Objective radiographic staging with a) contrast-enhanced, helical thin-cut computed tomography (CT)/magnetic resonance imaging (MRI) scan of the abdomen and b) CT scan/MRI of the chest
  * Note: echoendoscopic staging will be permitted as an adjunctive modality, but all stage definitions below will be determined using CT/MRI as outlined below. In the event echoendoscopic stage and CT/MRI stage are discordant, the CT/MRI stage will be used. Significant discordance should be discussed with the study principal investigator (PI) prior to enrollment
  * Borderline resectable primary tumor, defined by the presence of any one or more of the following on CT/MRI, and confirmed by central radiographic review:

    * An interface between the primary tumor and the superior mesenteric vein or portal vein (SMV-PV) measuring ≥ 180 degrees of the circumference of the vessel wall
    * Short-segment occlusion of the SMV-PV with normal vein above and below the level of obstruction that is amenable to resection and venous reconstruction
    * Short segment interface (of any degree) between tumor and hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and reconstruction
    * An interface between the tumor and superior mesenteric artery (SMA) measuring < 180 degrees of the circumference of the vessel wall
  * No potentially resectable disease defined as primary tumors with all of the following:

    * An interface between the primary tumor and the superior mesenteric vein or portal vein (SMV-PV) measuring < 180 degrees of the circumference of the vessel wall
    * No radiographic interface between the tumor and the (superior mesenteric artery) SMA, hepatic artery or celiac axis
    * No radiographic evidence of metastatic disease
  * No metastatic disease defined as any one or more of the following:

    * Suspicious lymphadenopathy outside the standard surgical field (i.e., aortocaval nodes, distant abdominal nodes)
    * Radiographic evidence for metastatic disease in distant organs, such as masses in distant organs or ascites
  * No locally advanced and/or unresectable disease clearly defined by any one or more of the following by CT/MRI:

    * An interface between the tumor and the SMA measuring ≥ 180 degrees of the circumference of the vessel wall
    * No interface between the tumor and the aorta
    * Occlusion of the SMV or portal vein without a sufficient cuff of normal vein above and below the level of obstruction with which to perform venous reconstruction
    * Long-segment interface (of any degree) between the tumor and the common hepatic artery or its major tributaries with insufficient artery proximal and distal to the interface to perform reconstruction
* No prior chemotherapy or chemoradiation for pancreatic cancer
* No patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years
* Baseline peripheral sensory neuropathy must be grade < 2
* No patients with known Gilbert's Syndrome or homozygosity for UGT1A1*28 polymorphism
* No history of pulmonary embolism in the past 6 months
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status 0-1
* Pregnancy/Nursing Status: Non-pregnant and non-breast-feeding. Female participants of child-bearing potential must have a negative urine or serum pregnancy test prior to registration. Perimenopausal participants must be amenorrheic > 12 months to be considered not of childbearing potential.
* Required Pre-Registration Laboratory Values:

  * Granulocytes ≥ 2,000/ul
  * Hemoglobin > 9 g/dL
  * Platelets ≥ 100,000/ul
  * Albumin > 3.0 g/dL
  * Creatinine ≤1.5 x upper limit of normal (ULN)

Registration Eligibility Criteria

* Confirmation of pre-registration eligibility criteria as described under "Documentation of Disease and Radiographic Staging" by the Alliance Central Radiographic Review
* Required Registration Laboratory Values:

  * Bilirubin ≤2 mg/dl
  * AST (SGOT) & ALT (SGPT) ≤ 2.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Accrual rate, calculated by total number of patients accrued divided by number of months from the date the study is opened at the fifth site to the evaluation date | Up to 3 years
Rate of treatment-related toxicity during preoperative therapy assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4 | Up to 30 days after completion of study treatment
Rate of treatment delay (greater than 4 weeks) during preoperative therapy | Up to 28 weeks
Completion rate of all preoperative and operative therapy | Up to 30 weeks

SECONDARY OUTCOMES:
Macroscopic (R0/R1) resection rate defined as number of patients achieved R0 or R1 resection during surgery divided by number of evaluable patients | At the time of surgery
Radiographic response rate defined as number of patients who achieved complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 during pre-operative therapy divided by the number of evaluable patients | Up to 18 weeks
Histopathologic response rate defined as number of patients who achieved CR or PR determined according to histopathologic examination during pre-operative therapy divided by the number of evaluable patients | Up to 18 weeks
Time to locoregional recurrence | From the date of registration to the date of the first documented locoregional recurrence, assessed up to 3 years
Time to distant recurrence | From the date of registration to the date of the first documented distant recurrence, assessed up to 3 years
Overall survival | From the date of registration to the date of the death due to all causes, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Katz, M.D., Study Chair — M.D. Anderson Cancer Center
Locations (14):
- United States (14):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University Pointe, West Chester, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Katz MH, Shi Q, Ahmad SA, Herman JM, Marsh Rde W, Collisson E, Schwartz L, Frankel W, Martin R, Conway W, Truty M, Kindler H, Lowy AM, Bekaii-Saab T, Philip P, Talamonti M, Cardin D, LoConte N, Shen P, Hoffman JP, Venook AP. Preoperative Modified FOLFIRINOX Treatment Followed by Capecitabine-Based Chemoradiation for Borderline Resectable Pancreatic Cancer: Alliance for Clinical Trials in Oncology Trial A021101. JAMA Surg. 2016 Aug 17;151(8):e161137. doi: 10.1001/jamasurg.2016.1137. Epub 2016 Aug 17. PMID 27275632